CLINICAL TRIAL: NCT07367048
Title: The Effect of the Four Life Domains Vision Board Program on Hope and Psychological Resilience in Adolescents Undergoing Cancer Treatment: A Randomized Controlled Trial
Brief Title: Four Life Domains Vision Board Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hazal Ozdemir Koyu, Dr. Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2026-65
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Children With Cancer
Keywords: adolescent cancer; Vision board intervention; hope; Psychosocial intervention

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel-group randomized controlled trial. Eligible adolescents undergoing cancer treatment will be randomly assigned to either the intervention group or the control group in a 1:1 ratio. The intervention group will receive a structured five-week Vision Board Program based on four life domains (health, well-being, love, and self-expression), while the control group will continue to receive standard hospital care without any additional psychosocial intervention. Outcomes will be assessed at baseline (pre-intervention) and after completion of the intervention (post-intervention). Outcome assessors will be blinded to group allocation due to the nature of the study.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. Due to the nature of the psychosocial intervention, participants and intervention providers cannot be blinded to group assignment. However, outcome assessors and data analysts will be blinded to group allocation to minimize assessment bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Received standart care
- Four Life Domains Vision Board Program (Experimental): Received Four Life Domains Vision Board Program
  Interventions: Other: Four Life Domains Vision Board Program

INTERVENTIONS:
Other: Four Life Domains Vision Board Program — The Four Life Domains-Based Vision Board Program is a structured psychosocial intervention designed to enhance hope and psychological resilience in adolescents undergoing cancer treatment. The program is grounded in positive psychology, mindfulness, and expressive arts approaches and focuses on four core life domains: health, well-being, love/relationships, and self-expression.
  The intervention consists of five weekly sessions (four core modules and one reinforcement session), delivered once per week. Each session includes guided breathing exercises, mindfulness-based awareness practices, and creative art activities centered on vision board development. Adolescents actively create and expand a personalized vision board throughout the program by adding visual, symbolic, and written elements reflecting personal strengths, goals, values, emotional resources, and future-oriented hopes within each life domain.
  Session modules include: (1) Breath and First Light: Opening the Door to Self, f
  Arms: Four Life Domains Vision Board Program

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a Four Life Domains-Based Vision Board Program on hope and psychological resilience among adolescents undergoing cancer treatment. Adolescents receiving cancer treatment often experience psychological distress that may negatively affect their sense of hope and resilience. Vision board-based psychosocial interventions grounded in positive psychology and creative expression may support adaptive coping and emotional well-being.

The study will be conducted in pediatric hematology-oncology units of Gazi University Health Application and Research Center and Etlik City Hospital in Türkiye. A total of 60 adolescents aged 12-18 years who have been receiving cancer treatment for at least six months will be randomly assigned to either the intervention group (n=30) or the control group (n=30).

Participants in the intervention group will receive a structured 5-week Four Life Domains-Based Vision Board Program, consisting of four core modules and one reinforcement session, while the control group will receive standard hospital care only. Outcome measures, including hope and psychological resilience, will be assessed at baseline and after completion of the intervention. The findings are expected to contribute to the development of innovative and holistic psychosocial support interventions for adolescents undergoing cancer treatment.

DETAILED DESCRIPTION:
This study is designed as a parallel-group randomized controlled trial to evaluate the effectiveness of a Four Life Domains-Based Vision Board Program on hope and psychological resilience in adolescents undergoing cancer treatment. Adolescents receiving cancer therapy are exposed to prolonged physical symptoms and psychosocial stressors, which may negatively impact emotional well-being, hope, and resilience. Therefore, supportive psychosocial interventions that promote self-expression, meaning-making, and positive future orientation are needed.

The study will be conducted in the pediatric hematology-oncology units of Gazi University Health Application and Research Center and Etlik City Hospital in Türkiye during 2026. The study population will consist of adolescents aged 12-18 years who have been receiving cancer treatment for at least six months. A total of 60 participants will be enrolled, with 30 adolescents allocated to the intervention group and 30 to the control group.

Participants meeting the inclusion criteria will be assigned a unique study identification number. Stratified block randomization based on age and gender will be applied. Random allocation will be performed by an independent statistician using a computerized randomization tool, and group assignments will be concealed in sealed, opaque envelopes to ensure allocation concealment.

The intervention group will participate in a structured Five-Week Vision Board Program grounded in four life domains: health, well-being, love/connection, and self-expression. The program includes weekly sessions integrating guided breathing exercises, mindfulness practices, creative art-based activities, and vision board creation processes. The modules include:

Breath and First Light: Opening the Door to Self

My Potential and Resources: Mapping My Strengths

Connection and Love: My Circle of Heart

Self-Expression: My Story and My Future

Reinforcement Session: The Big Picture - Reframing Hope

During each session, participants will progressively add visual and symbolic elements to their personal vision boards. The final session focuses on integrating the vision board as a holistic representation of hope and resilience.

The control group will receive standard hospital care without any additional psychosocial intervention. Data will be collected using a Sociodemographic Information Form, the Hope Scale for Adolescents, and the Psychological Resilience Scale. Assessments will be conducted at baseline (pre-test) and after completion of the five-week intervention (post-test). When necessary, data collection tools will be administered electronically via secure online platforms.

The effectiveness of the intervention will be evaluated by comparing pre- and post-intervention changes in hope and psychological resilience between the intervention and control groups. This study aims to provide evidence for a feasible, creative, and holistic psychosocial support model for adolescents undergoing cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18
* Has been receiving cancer treatment for at least 6 months
* Able to communicate in Turkish
* Not in the terminal stage

Exclusion Criteria:

* Those who have experienced a serious traumatic life event in the last 6 months
* Those with a psychiatric diagnosis
* Those with a medical condition that would prevent participation in the intervention

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Adolescent Hopefulness Scale, | Baseline (pre-intervention) and immediately after completion of the 5-week intervention
  Hope level will be assessed using the Adolescent Hopefulness Scale, a 24-item visual analog scale developed by Hinds and Gattuso and validated for Turkish adolescents aged 12-18 years. The scale measures adolescents' positive future expectations and hope at the time of assessment. Each item is scored on a 100-mm visual analog line, with total scores ranging from 0 to 2400. Higher scores indicate higher levels of hope.
Psychological Resilience | Baseline (pre-intervention) and immediately after completion of the 5-week intervention
  Psychological resilience will be measured using the Child and Youth Resilience Measure (CYRM-28), which assesses individual, relational, and contextual resilience resources in adolescents aged 12-18 years. The scale consists of 28 items rated on a 5-point Likert scale. Higher total scores indicate greater psychological resilience.

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data has not yet been made. Any future data sharing will be considered following completion of the study, in accordance with ethical approval, participant consent, and applicable data protection regulations.

REFERENCES:
- [Result] 1. Esenay FI, Conk Z. Ergenler için Umutluluk Ölçeği: Geçerlik-güvenirlik çalışması.(2012). Ankara Sağlık Bilimleri Dergisi, 2, 230-248. 2. Arslan, G. (2015). Ergenlerde psikolojik sağlamlık: Bireysel koruyucu faktörlerin rolü. Türk Psikolojik Danışma ve Rehberlik Dergisi, 5(44), 149-158. 3. Ball, J., Bindler, R. M., Cowen, K. J., & Shaw, M. R. (2017). Principles of pediatric nursing : caring for children (Seventh ed.). Pearson Education. 4. Dupuis, L. L., Vettese, E., Aftandilian, C., Agarwal, V., Baggott, C., Bradfield, S. M., Crellin-Parsons, N., Freyer, D. R., Kelly, K. M., & King, A. A. (2025). Factors Associated With Self-Report Symptom Screening Adherence in Pediatric Cancer Patients. Cancer Medicine, 14(14), e71053. 5. Jin, X., Li, H., Chong, Y. Y., Mann, K. F., Yao, W., & Wong, C. L. (2023). Feasibility and preliminary effects of acceptance and commitment therapy on reducing psychological distress and improving the quality of life of the parents of children with cancer: A pilot randomised controlled trial. Psycho-oncology, 32(1), 165-169. 6. Kisecik Sengul, Z., & Kilicarslan, E. (2025). Investigation into the impact of technology-based motivation program applied to children following cancer diagnosis and their families: a randomized controlled study. BMC psychology, 13(1), 857. 7. O'Daffer, A., Comiskey, L., Scott, S. R., Zhou, C., Bradford, M. C., Yi-Frazier, J. P., & Rosenberg, A. R. (2023). Protocol for the promoting resilience in stress management (PRISM) intervention: a multi-site randomized controlled trial for adolescents and young adults with advanced cancer. BMC Palliative Care, 22(1), 1-9. 8. Ozdemir Koyu, H., & Tas Arslan, F. (2021). The effect of physical and psychosocial symptoms on caregiver burden of parents of children with cancer. European Journal of Cancer Care, 30(6), e13513. 9. Tutelman, P. R., Moran, C., Beattie, S. M., Khu, M., Howlett, M., Scheidl, J., Boychuk, A., Silveira, K., Henning, J. W., & Schulte, F. S. (2024). Acceptab